CLINICAL TRIAL: NCT04546360
Title: Spleen Stiffness Combined With Liver Stiffness Measured by Two-dimensional Shear Wave Elastography for the Screening of High-risk Varices in Patients With Compensated Advanced Chronic Liver Disease (CHESS2004)
Brief Title: Spleen Stiffness Combined With Liver Stiffness Measured by 2D-SWE for the Screening of High-risk Varices in Compensated Advanced Chronic Liver Disease (CHESS2004)
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Tianjin Second People's Hospital (Other); The Sixth People's Hospital of Shenyang (Other); Hospital of the Chengdu Office of the People's Government of Tibet Autonomous Region (Unknown); The Central Hospital of Lishui City (Other); Guangxi Zhuang Autonomous Region (Unknown)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2004
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Compensated Advanced Chronic Liver Disease; Variceal Hemorrhage
Keywords: Spleen stiffness; Liver stiffness; Two-dimensional shear wave elastography; High-risk varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants will receive standard esophagogasrtoduodendoscopy, spleen stiffness measurement and liver stiffness measurement based on two-dimensional shear wave elastography, gallbladder wall thickness, spleen thickness, spleen long diameter and serological examination (platelet count, alanine aminotransferase, aspartate aminotransferase, total bilirubin, creatinine, albumin, prothrombin time, international normalized ratio).
  Interventions: Procedure: Esophagogasrtoduodendoscopy, spleen stiffness measurement and liver stiffness measurement.

INTERVENTIONS:
Procedure: Esophagogasrtoduodendoscopy, spleen stiffness measurement and liver stiffness measurement. — Time frame between elastography measurement and esophagogastroduodendoscopy is within 2 weeks.

SUMMARY:
Variceal hemorrhage is the serious complication in patients with compensated advanced chronic liver disease (cACLD). To evaluate the bleeding risk of varices, esophagogastroduodenoscopy (EGD) should be performed. However, EGD is limited by its invasiveness and uncomfortableness. The Baveno VI criteria recommended that EGD could be spared in patients with liver stiffness (LS) based on transient elastography (TE) < 20 kPa and platelet count >150000/mm3. However, only 30% of patients can spare EGD. In order to expand the screening criteria, Expanded-Baveno VI proposed that by using LS (TE)<25 kPa and platelet count >110000/mm3, 40% of patients can safely avoid EGD. It is worth noting that the Baveno VI criteria is based on the European and American compensatory cirrhosis cohort (55% for hepatitis C, 14% for non-alcoholic steatohepatitis, 13% for alcoholic hepatitis, 8% for hepatitis B), Expanded-Baveno VI is also of good diagnostic value for hepatitis C, alcoholic, and non-alcoholic steatohepatitis of cACLD. About 257 million people worldwide are infected with hepatitis B virus, and about 80 million people in China alone are infected with hepatitis B virus. Infected with hepatitis B virus is the main etiology of patients with cACLD in china. Hence, Baveno VI and Expanded-Baveno VI may not be suitable for patients with hepatitis B virus-dominant cACLD.

Previous studies have shown that LS has a significant correlation with the severity of portal hypertension. Nevertheless, LS only has a good correlation with portal pressure in the early stage of portal hypertension (hepatic vein pressure gradient ≤10mm Hg), because liver fibrosis is the main cause of portal hypertension in this period. In the late stage of liver cirrhosis, the involvement of hyperdynamic circulation and increased portal blood flow, spleen stiffness (SS) may have a better correlation with HVPG than that of LS. Therefore, SS provides a reliable basis for the hemodynamic changes that occur during the development of liver cirrhosis and avoids the limitations caused by the measurement of LS. Previous study has found that changes in SS before and after non-selective beta-blockers (NSBBs) as primary prophylaxis may be a promising non-invasive tool for predicting hemodynamic response in patients with high-risk varices.

Since SS is much higher than LS, the maximum threshold of 75 kPa measured with TE may not be sufficient to evaluate the hardness of the spleen. Meanwhile, numerous studies have found that the success rate of measuring SS and LS based on 2D-SWE is higher than that of TE. Hence, CHESS2004 study aims to establish a standard for predicting high-risk varices that is more suitable in patients with hepatitis B virus-dominant cACLD. In addition, non-invasive means of SS is used to evaluate the hemodynamic response of patients with high-risk varices receiving prophylaxis NSBBs therapy.

DETAILED DESCRIPTION:
Variceal hemorrhage is the serious complication in patients with compensated advanced chronic liver disease (cACLD). To evaluate the bleeding risk of varices, esophagogastroduodenoscopy (EGD) should be performed. However, EGD is limited by its invasiveness and uncomfortableness. The Baveno VI criteria recommended that EGD could be spared in patients with liver stiffness (LS) based on transient elastography (TE) < 20 kPa and platelet count >150000/mm3. However, only 30% of patients can spare EGD. In order to expand the screening criteria, Expanded-Baveno VI proposed that by using LS (TE)<25 kPa and platelet count >110000/mm3, 40% of patients can safely avoid EGD. It is worth noting that the Baveno VI criteria is based on the European and American compensatory cirrhosis cohort (55% for hepatitis C, 14% for non-alcoholic steatohepatitis, 13% for alcoholic hepatitis, 8% for hepatitis B), Expanded-Baveno VI is also of good diagnostic value for hepatitis C, alcoholic, and non-alcoholic steatohepatitis of cACLD. About 257 million people worldwide are infected with hepatitis B virus, and about 80 million people in China alone are infected with hepatitis B virus. Infected with hepatitis B virus is the main etiology of patients with cACLD in china. Hence, Baveno VI and Expanded-Baveno VI may not be suitable for patients with hepatitis B virus-dominant cACLD.

Previous studies have shown that LS has a significant correlation with the severity of portal hypertension. Nevertheless, LS only has a good correlation with portal pressure in the early stage of portal hypertension (hepatic vein pressure gradient ≤10mm Hg), because liver fibrosis is the main cause of portal hypertension in this period. In the late stage of liver cirrhosis, the involvement of hyperdynamic circulation and increased portal blood flow, spleen stiffness (SS) may have a better correlation with HVPG than that of LS. Therefore, SS provides a reliable basis for the hemodynamic changes that occur during the development of liver cirrhosis and avoids the limitations caused by the measurement of LS. Previous study has found that changes in SS before and after non-selective beta-blockers (NSBBs) as primary prophylaxis may be a promising non-invasive tool for predicting hemodynamic response in patients with high-risk varices.

Since SS is much higher than LS, the maximum threshold of 75 kPa measured with TE may not be sufficient to evaluate the hardness of the spleen. Numerous studies have found that the success rate of measuring SS and LS based on two-dimensional shear wave elastography is higher than that of TE. Hence, CHESS2004 study in seven centers including LanZhou University, Tianjin Second People's Hospital, Sixth People's Hospital of Shenyang, Hospital of the Chengdu Office of the People's Government of Tibet Autonomous Region, The Central Hospital of Lishui City and Guangxi Zhuang Autonomous Region, aims to establish a standard for predicting high-risk varices that is more suitable in patients with hepatitis B virus-dominant cACLD. In addition, non-invasive means of SS is used to evaluate the hemodynamic response of patients with high-risk varices receiving prophylaxis NSBBs therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* confirmed cirrhosis based on liver biopsy or clinical findings;
* without decompensated events (e.g. ascites, bleeding, or overt encephalopathy);
* scheduled to undergo esophagogastroduodenoscopy, spleen stiffness measurement and liver stiffness measurement;
* estimated survival time>24 months, and model for end-stage liver disease score<19, and without liver transplant;
* with written informed consent.

Exclusion Criteria:

* contradictions for esophagogastroduodenoscopy;
* accepted primary prevention (non-selective beta blockers or endoscopic variceal ligation);
* time frame between elastography measurement and esophagogastroduodenoscopy>14 days;
* diagnosed as hepatocellular carcinoma;
* absence of spleen or splenectomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with compensated advanced chronic liver disease
Sampling Method: Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of combined model of spleen stiffness and liver stiffness | 1 day
  To assess the accuracy of combined model of spleen stiffness and liver stiffness to avoid unnecessary esophagogasrtoduodendoscopy in patients with compensated advanced chronic liver disease

SECONDARY OUTCOMES:
Accuracy of LSPS model base on two-dimensional shear wave elastography | 1 day
  To assess the accuracy of LSPS (liver stiffness-spleen size- to platelet ration risk score) base on two-dimensional shear wave elastography for high-risk varices in patients with compensated advanced chronic liver disease
Rate of hemodynamic responder of patients receiving prophylaxis NSBBs therapy | 1 month
  Rate of hemodynamic responder of patients receiving prophylaxis NSBBs therapy assessed by spleen stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, MD, Study Chair — LanZhou University; Linxue Qian, MD, Study Chair — Beijing Friendship Hospital; Fengmei Wang, MD, Principal Investigator — Tianjin Second People's Hospital; Ye Gu, MD, Principal Investigator — The Sixth People's Hospital of Shenyang; Chao Liu, MD, Principal Investigator — Hospital of the Chengdu Office of the People's Government of Tibet Autonomous Region; Chuxiao Shao, MD, Principal Investigator — The Central Hospital of Lishui City; Guo Zhang, MD, Principal Investigator — Guangxi Zhuang Autonomous Region; Sumei Ma, MD, Principal Investigator — LanZhou University
Locations (6):
- China (6):
  - Guangxi Zhuang Autonomous Region, Guangxi
  - Lanzhou University, Lanzhou
  - The Central Hospital of Lishui City, Lishui
  - Sixth People's Hospital of Shenyang, Shenyang
  - Tianjin Second People's Hospital, Tianjin
  - Hospital of the Chengdu Office of the People's Government of Tibet Autonomous Region, Xi'zang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Maurice JB, Brodkin E, Arnold F, Navaratnam A, Paine H, Khawar S, Dhar A, Patch D, O'Beirne J, Mookerjee R, Pinzani M, Tsochatzis E, Westbrook RH. Validation of the Baveno VI criteria to identify low risk cirrhotic patients not requiring endoscopic surveillance for varices. J Hepatol. 2016 Nov;65(5):899-905. doi: 10.1016/j.jhep.2016.06.021. Epub 2016 Jul 5. PMID 27388923
- [Background] Augustin S, Pons M, Maurice JB, Bureau C, Stefanescu H, Ney M, Blasco H, Procopet B, Tsochatzis E, Westbrook RH, Bosch J, Berzigotti A, Abraldes JG, Genesca J. Expanding the Baveno VI criteria for the screening of varices in patients with compensated advanced chronic liver disease. Hepatology. 2017 Dec;66(6):1980-1988. doi: 10.1002/hep.29363. Epub 2017 Oct 30. PMID 28696510
- [Background] Hirooka M, Ochi H, Koizumi Y, Kisaka Y, Abe M, Ikeda Y, Matsuura B, Hiasa Y, Onji M. Splenic elasticity measured with real-time tissue elastography is a marker of portal hypertension. Radiology. 2011 Dec;261(3):960-8. doi: 10.1148/radiol.11110156. Epub 2011 Sep 16. PMID 21926379
- [Background] Cooke GS, Andrieux-Meyer I, Applegate TL, Atun R, Burry JR, Cheinquer H, Dusheiko G, Feld JJ, Gore C, Griswold MG, Hamid S, Hellard ME, Hou J, Howell J, Jia J, Kravchenko N, Lazarus JV, Lemoine M, Lesi OA, Maistat L, McMahon BJ, Razavi H, Roberts T, Simmons B, Sonderup MW, Spearman CW, Taylor BE, Thomas DL, Waked I, Ward JW, Wiktor SZ; Lancet Gastroenterology & Hepatology Commissioners. Accelerating the elimination of viral hepatitis: a Lancet Gastroenterology & Hepatology Commission. Lancet Gastroenterol Hepatol. 2019 Feb;4(2):135-184. doi: 10.1016/S2468-1253(18)30270-X. PMID 30647010
- [Background] Kim HY, So YH, Kim W, Ahn DW, Jung YJ, Woo H, Kim D, Kim MY, Baik SK. Non-invasive response prediction in prophylactic carvedilol therapy for cirrhotic patients with esophageal varices. J Hepatol. 2019 Mar;70(3):412-422. doi: 10.1016/j.jhep.2018.10.018. Epub 2018 Oct 31. PMID 30389550